CLINICAL TRIAL: NCT07322133
Title: Dopamine vs. Norepinephrine in Term and Late Preterm Neonates With Hypoxemic Respiratory Failure and Systemic Hypotension Due to Pulmonary Hypertension: A Pilot Trial
Brief Title: Dopamine vs. Norepinephrine for Hypotension in Neonates With Pulmonary Hypertension (DONE)
Acronym: DONE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Children's Miracle Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2339428; GFDS25 (Other Grant/Funding Number: Children's Miracle Network Research Grant)
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hypotension and Shock; Pulmonary Hypertension of the Newborn (PPHN); Hypoxemic Respiratory Failure
Keywords: Pulmonary Hypertension; Systemic Hypotension; Vasopressor
MeSH Terms: conditions — Hypotension; Shock; Respiratory Insufficiency; Hypertension, Pulmonary | interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dopamine Arm (Active Comparator): Infants in this group will receive dopamine as their first-line vasopressor. Continuous intravenous dopamine infusion will be initiated at 5 mcg/kg/min and titrated to achieve gestational age appropriate mean arterial blood pressure targets (maximum 20 mcg/kg/min).
  Interventions: Drug: Dopamine administration
- Norepinephrine Arm (Active Comparator): Infants in this group will receive norepinephrine as their first-line vasopressor. Continuous intravenous norepinephrine infusion initiated at 0.02 mcg/kg/min and titrated to achieve gestational age appropriate mean arterial blood pressure targets (maximum 1 mcg/kg/min).
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Dopamine administration — Infants meeting the inclusion criteria who are randomized to dopamine arm will receive dopamine infusion starting at 5 mcg/kg/min, titrated to mean arterial pressure targets based on gestational age, max dose 20 mcg/kg/min.
  Arms: Dopamine Arm
Drug: Norepinephrine — Infants meeting the inclusion criteria who are randomized to norepinephrine arm will receive norepinephrine infusion starting at 0.02 mcg/kg/min, titrated to mean arterial pressure targets based on gestational age, max dose 1 mcg/kg/min.
  Arms: Norepinephrine Arm

SUMMARY:
This pilot randomized clinical trial compares dopamine and norepinephrine as first-line vasoactive therapies in term and late preterm neonates with pulmonary hypertension associated with hypoxemic respiratory failure and systemic hypotension. Systemic hypotension is a common and clinically significant complication of persistent pulmonary hypertension of the newborn (PPHN) and frequently requires vasopressor support to maintain adequate systemic perfusion. Dopamine is commonly used in this setting; however, prior animal experimental and clinical data suggest it may increase pulmonary vascular resistance, potentially worsening right ventricular afterload and hypoxemia. Norepinephrine may preferentially increase systemic vascular resistance with less effect on the pulmonary circulation. This study evaluates short-term hemodynamic and oxygenation responses following initiation of dopamine or norepinephrine.

DETAILED DESCRIPTION:
Persistent pulmonary hypertension of the newborn (PPHN) is a serious cardiopulmonary disorder characterized by sustained elevation of pulmonary vascular resistance, leading to right-to-left shunting, impaired oxygenation, and increased morbidity and mortality. In addition to hypoxemic respiratory failure, many infants with PPHN develop systemic hypotension. Management of systemic hypotension in this population is complex, as vasoactive medications may have differing effects on systemic and pulmonary circulations.

Dopamine is widely used as first-line therapy for neonatal hypotension because of its dose-dependent dopaminergic and adrenergic effects. However, both animal models and clinical observations suggest that dopamine may increase pulmonary vascular resistance in neonates with PPHN. Norepinephrine, a predominantly alpha-adrenergic agonist with modest beta-adrenergic activity, may provide more selective augmentation of systemic vascular resistance while exerting less influence on pulmonary vascular tone. Despite the increasing clinical use of norepinephrine in neonatal intensive care units, there are no prospective trials comparing dopamine and norepinephrine in neonates with PPHN.

This is a single-center, cluster-randomized, pilot clinical trial enrolling term and late preterm neonates with hypoxemic respiratory failure, echocardiographic evidence of pulmonary hypertension, and systemic hypotension that persists despite initial fluid resuscitation. Eligible infants are assigned by time-based cluster randomization to receive either dopamine or norepinephrine as first-line vasoactive therapy, consistent with standard clinical practice in the neonatal intensive care unit. Informed consent is obtained for research-specific procedures, including serial targeted neonatal echocardiography, while vasoactive medication use follows established clinical protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenstrual age > 34 6/7 weeks and Postnatal age ≤ 28 days
2. On respiratory support (Invasive mechanical ventilation, NIPPV, CPAP, HFNC ≥ 2 LPM) and FiO2 ≥ 0.3
3. Echocardiographic evidence of pulmonary hypertension
4. Mean arterial pressure below the threshold for gestational age despite a 10-20 mL/kg fluid bolus

Permissible Comorbidities: CDH, trisomy 21, HIE on hypothermia, PDA, PFO/ASD, VSD < 2 mm

Exclusion Criteria:

1. Gestational age < 32 weeks
2. Severe hypoxic respiratory failure (OI > 35 or SpO2 < 75% on 100% FiO2 for > 60 minutes)
3. Lethal anomalies (e.g., trisomy 13 or 18)
4. Complex congenital heart disease beyond specified criteria

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
SAP/PAP ratio | Within 30 hours of vasopressor initiation.
  Ratio of systemic arterial pressure to pulmonary arterial pressure (SAP/PAP)
LV Cardiac output | Within 30 hours of vasopressor initiation
  Left Ventricular Cardiac Output calculated with echocardiography
Oxygenation Indices | Within 30 hours of vasopressor initiation
  FiO₂ (fraction of inspired oxygen), SpO₂ (peripheral oxygen saturation), PaO₂ (arterial oxygen partial pressure), OI (oxygenation index), OSI (oxygen saturation index)

SECONDARY OUTCOMES:
Use of inhaled nitric oxide (iNO) | Within 30 hours of vasopressor initiation
Need for additional vasoactive agents | Within 30 hours of vasopressor initiation
Echocardiographic markers of heart function | Within 30 hours of vasopressor initiation
  Right ventricle and Left ventricle function

CONTACTS AND LOCATIONS:
Overall Officials: Deepika Sankaran, MD, Principal Investigator — UC Davis Health
Locations (1):
- UC Davis Children's Hospital, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jain A, El-Khuffash AF, van Herpen CH, Resende MHF, Giesinger RE, Weisz D, Mertens L, Jankov RP, McNamara PJ. Cardiac Function and Ventricular Interactions in Persistent Pulmonary Hypertension of the Newborn. Pediatr Crit Care Med. 2021 Feb 1;22(2):e145-e157. doi: 10.1097/PCC.0000000000002579. PMID 33044416
- [Background] Lesneski AL, Vali P, Hardie ME, Lakshminrusimha S, Sankaran D. Randomized Trial of Oxygen Saturation Targets during and after Resuscitation and Reversal of Ductal Flow in an Ovine Model of Meconium Aspiration and Pulmonary Hypertension. Children (Basel). 2021 Jul 14;8(7):594. doi: 10.3390/children8070594. PMID 34356574
- [Background] Siefkes HM, Lakshminrusimha S. Management of systemic hypotension in term infants with persistent pulmonary hypertension of the newborn: an illustrated review. Arch Dis Child Fetal Neonatal Ed. 2021 Jul;106(4):446-455. doi: 10.1136/archdischild-2020-319705. Epub 2021 Jan 21. PMID 33478959
- [Background] Lakshminrusimha S. The pulmonary circulation in neonatal respiratory failure. Clin Perinatol. 2012 Sep;39(3):655-83. doi: 10.1016/j.clp.2012.06.006. PMID 22954275
- [Background] Tourneux P, Rakza T, Bouissou A, Krim G, Storme L. Pulmonary circulatory effects of norepinephrine in newborn infants with persistent pulmonary hypertension. J Pediatr. 2008 Sep;153(3):345-9. doi: 10.1016/j.jpeds.2008.03.007. Epub 2008 May 12. PMID 18534241
- [Background] Steinhorn RH. Neonatal pulmonary hypertension. Pediatr Crit Care Med. 2010 Mar;11(2 Suppl):S79-84. doi: 10.1097/PCC.0b013e3181c76cdc. PMID 20216169
- [Background] Sankaran D, Lakshminrusimha S. Pulmonary hypertension in the newborn- etiology and pathogenesis. Semin Fetal Neonatal Med. 2022 Aug;27(4):101381. doi: 10.1016/j.siny.2022.101381. Epub 2022 Aug 7. PMID 35963740
- [Background] McNamara PJ, Giesinger RE, Lakshminrusimha S. Dopamine and Neonatal Pulmonary Hypertension-Pressing Need for a Better Pressor? J Pediatr. 2022 Jul;246:242-250. doi: 10.1016/j.jpeds.2022.03.022. Epub 2022 Mar 18. No abstract available. PMID 35314154
- [Background] Liet JM, Boscher C, Gras-Leguen C, Gournay V, Debillon T, Roze JC. Dopamine effects on pulmonary artery pressure in hypotensive preterm infants with patent ductus arteriosus. J Pediatr. 2002 Mar;140(3):373-5. doi: 10.1067/mpd.2002.123100. PMID 11953739
- [Background] Cheung PY, Barrington KJ. The effects of dopamine and epinephrine on hemodynamics and oxygen metabolism in hypoxic anesthetized piglets. Crit Care. 2001;5(3):158-66. doi: 10.1186/cc1016. Epub 2001 Apr 26. PMID 11353933
- [Background] Budniok T, ElSayed Y, Louis D. Effect of Vasopressin on Systemic and Pulmonary Hemodynamics in Neonates. Am J Perinatol. 2021 Oct;38(12):1330-1334. doi: 10.1055/s-0040-1712999. Epub 2020 Jun 2. PMID 32485754
- [Background] Shah S, Dhalait S, Fursule A, Khandare J, Kaul A. Use of Vasopressin as Rescue Therapy in Refractory Hypoxia and Refractory Systemic Hypotension in Term Neonates with Severe Persistent Pulmonary Hypertension-A Prospective Observational Study. Am J Perinatol. 2024 May;41(S 01):e886-e892. doi: 10.1055/a-1969-1119. Epub 2022 Oct 27. PMID 36302521
- [Background] McNamara PJ, Jain A, El-Khuffash A, Giesinger R, Weisz D, Freud L, Levy PT, Bhombal S, de Boode W, Leone T, Richards B, Singh Y, Acevedo JM, Simpson J, Noori S, Lai WW. Guidelines and Recommendations for Targeted Neonatal Echocardiography and Cardiac Point-of-Care Ultrasound in the Neonatal Intensive Care Unit: An Update from the American Society of Echocardiography. J Am Soc Echocardiogr. 2024 Feb;37(2):171-215. doi: 10.1016/j.echo.2023.11.016. PMID 38309835
- [Background] de Boode WP, Singh Y, Gupta S, Austin T, Bohlin K, Dempsey E, Groves A, Eriksen BH, van Laere D, Molnar Z, Nestaas E, Rogerson S, Schubert U, Tissot C, van der Lee R, van Overmeire B, El-Khuffash A. Recommendations for neonatologist performed echocardiography in Europe: Consensus Statement endorsed by European Society for Paediatric Research (ESPR) and European Society for Neonatology (ESN). Pediatr Res. 2016 Oct;80(4):465-71. doi: 10.1038/pr.2016.126. Epub 2016 Jun 8. No abstract available. PMID 27384404